CLINICAL TRIAL: NCT01864954
Title: Web and Phone Intervention to Maintain Postpartum Tobacco Abstinence
Acronym: StayQuit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01CA140310-01A2 (NIH)
Record Dates: First submitted 2013-05-01; First posted 2013-05-30 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Smoking
Keywords: Smoking; Postpartum; Pregnancy; Quit; Tobacco; Abstinence; Relapse; Relapse prevention
MeSH Terms: conditions — Smoking; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Web+phone (Experimental): Engaging and interactive website access plus phone calls from personal coach.
  Interventions: Behavioral: Web+phone
- Basic Static Web (Active Comparator): Static website access only, only introductory call.
  Interventions: Behavioral: Web+phone

INTERVENTIONS:
Behavioral: Web+phone — We propose to evaluate the feasibility, acceptability, and efficacy of a Web+phone treatment program in a small, randomized, controlled pilot study. Women who have quit smoking during pregnancy will be randomly assigned to either (a) an Enhanced Web+phone intervention or (b) a Basic Web Information-Only control condition.

SUMMARY:
This study seeks to develop and test a Web-based tobacco relapse prevention program targeting postpartum women who quit smoking for pregnancy. Participants are randomly assigned to one of two conditions: (1) an Enhanced Web+phone Condition that receives access to an interactive Web-based intervention plus up to 3 brief supportive phone calls from a personal coach; (2) A Basic Web Information-Only Control Condition that receives access to an informational website plus an introductory phone call. The hypothesis is that Women in the Enhanced Condition will be more successful in avoiding tobacco relapse than women assigned to the Basic Control Condition.

DETAILED DESCRIPTION:
The primary aims of this project are to:

1. Adapt and refine an Enhanced Web+phone intervention for the maintenance of tobacco abstinence postpartum.
2. Evaluate the feasibility and acceptability of the Enhanced Web+phone tobacco abstinence maintenance program for postpartum women.

   Aim 2.1 The investigators hypothesize that the intervention will be feasible as assessed by women's report of helpfulness, relevance and program usability.

   Aim 2.2 The investigators hypothesize that the intervention will be acceptable to postpartum women as measured by engagement in and use of the program.
3. Estimate the initial efficacy of the Enhanced Web+phone intervention on tobacco abstinence at 3 and 6 months postpartum relative to a Basic Web Information-Only control.

Aim 3.1 The investigators hypothesize that, relative to the Basic Web Information-Only control, the Enhanced Web+phone intervention will be associated with 10-points greater prolonged abstinence rates at 3 and 6 months postpartum.

Aim 3.2 The investigators hypothesize that, relative to Basic Web control, tobacco use outcomes at 3 and 6 months postpartum in the Enhanced Web+phone intervention will be associated with greater improvements (d > .35) in putative mediators of prolonged abstinence (i.e., self-efficacy, intentions to maintain nonsmoking, mood and perceived stress, and weight concerns).

Secondary aim of this proposal is to:

Evaluate potential predictors of postpartum smoking relapse. The investigators will examine pre-pregnancy smoking rate, partner's tobacco use and other demographic factors as predictors of postpartum tobacco relapse. Similarly, the investigators will examine the role of mood, perceived stress and weight concerns as predictors of prolonged abstinence among women in both groups. For example, it may be that women with higher baseline levels of depressive symptoms and perceived stress may be more likely to return to smoking postpartum, regardless of condition.

ELIGIBILITY:
Inclusion Criteria:

* Smoked at least 5 cigarettes/day for at least 1 of the 3 months prior to becoming pregnant
* No smoking during weeks 34 to 38 of pregnancy
* Able to read English
* At least 18 years of age
* Use Web e-mail account at least once per week
* Completed informed assent/consent.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
All tobacco abstinence | 3 and 6 months postpartum
  Measure change in 7-day point all tobacco abstinence and change in prolonged abstinence between 3 and 6 months postpartum.

SECONDARY OUTCOMES:
Potential predictors of postpartum tobacco relapse | 6 months postpartum
  Measure change from baseline in participant-specific variables (e.g.,demographics, smoking history, partner tobacco use, mood, weight concerns) to examine possible predictors of postpartum tobacco relapse.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

REFERENCES:
- See also: Oregon Research Institute — http://www.ori.org